CLINICAL TRIAL: NCT06677216
Title: Botulinum Toxin in the Management of Temporo-mandibular Related Myalgia: a Prospective Study
Acronym: BOMAMY
Status: Enrolling by invitation | Type: Observational
Sponsor: Diakonessenhuis, Utrecht (Other)
Collaborators: Fysiotherapie Utrecht Oost B.V. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23-061; Wetenschapsbeurzen W2021-2001 (Other Grant/Funding Number: Onderzoeksfonds. St. Vrienden van het Diak)
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: TMD/Orofacial Pain; Myalgia of Mastication Muscle; Botulinum Toxin, Type a
Keywords: TMD; Myalgia; Orofacial pain; Botulinum Toxin A
MeSH Terms: conditions — Myalgia; Facial Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with TMD-related myalgia treated with BTX-A at the department of OMS: Participants for this study were adults with TMD-related myalgia according to the DC/TMD treated with a BTX-A injection. All participants were recruited at the department of Oral and Maxillofacial Surgery (OMS) of the Diakonessenhuis, Utrecht, The Netherlands.
  Interventions: Procedure: Botulinum Toxin, Type A

INTERVENTIONS:
Procedure: Botulinum Toxin, Type A — All participants will receive a solution of BTX-A (Xeomin, Merz Pharma GmbH, Frankfurt am Main, Germany) in the masseter and temporalis muscles (total of 100 units reconstituted with 4cc unpreserved 0.9% sodium chloride). The injection will be provided by the same maxillofacial surgeon. The participants are asked to clench their teeth to determine the site of the most intense muscle activity in the masseter and temporal muscles with palpation. Intramuscular BTX-A injections are administered on both sides at the location of the most intense muscle activity of the masseter (80 units) and temporalis (20 units).

SUMMARY:
The aim of this study was to evaluate the clinical course in terms of pain, function and quality of life of patients with TMD-related myalgia during six months after receiving BTX-A injections. The research question was: What are the outcomes in pain, quality of life and function of patients with TMD-related myalgia receiving BTX-A during 6 months? The hypothesis to be tested was that patients receiving a BTX-A injection due to TMD-related myalgia will have a reduction in pain and increase in quality of life and function after one, three- and six- months.

DETAILED DESCRIPTION:
This is a prospective and observational cohort study. The Medical Research Ethics Committees United provided a non-WMO (Medical Research Involving Human Subject Acts) waiver (W23.212) prior to commencement of this study. All participants will be informed and most give their written consent prior to participating, according the requirements of the Declaration of Helsinki (World Medical Association, 2013).

Participants Participants in this study are adults with TMD-related myalgia according to the DC/TMD treated with a BTX-A injection. All participants are recruited at the department of Oral and Maxillofacial Surgery (OMS) of the Diakonessenhuis, Utrecht, The Netherlands.

Inclusion criteria for participation are:

* TMD-related myalgia in accordance with the DC/TMD;
* Accepted BTX-A injections as treatment;
* Age ≥ 18 years;
* Understanding of the Dutch language to fill in the questionnaires.

Exclusion criteria for participation are:

* Systemic inflammatory and connective tissue diseases (e.g., rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis);
* Surgery in the TMJ area < 12 months ago;
* Pain of dental origin;
* Limited cognitive functioning (not allowed to make medical decisions);
* Use of muscle relaxants, or aminoglycoside antibiotics;
* A history of allergic reactions to BTX;
* Pregnancy and lactation.

Study procedure Participants willing to enroll in the study will recieve an information letter. After receiving all information participants will have two weeks to consider participation. When willing to participate they can contact the researcher for an appointment to sign the informed consent form and check for the inclusion/exclusion criteria.

During the first visit, participants will fill in their demographics, health history, previous treatments concerning TMD-related myalgia and presentation of current symptoms on a standard form. The researcher will check the presence of a TMD-related myalgia according to the DC/TMD.

Prior to the BTX-A injection, participants rate their pain on a Visual Analogue Scale (VAS). Next, the Oral Health Impact Profile-14 (OHIP-14) and the Mandibular Function Impairment Questionnaire (MFIQ) were administered. Then, the researcher will measure the maximum active and passive mouth opening according to the Dutch translation of the DC/TMD.

BTX-A injections All participants will recieve a solution of BTX-A (Xeomin, Merz Pharma GmbH, Frankfurt am Main, Germany) in the masseter and temporalis muscles (total of 100 units reconstituted with 4cc unpreserved 0.9% sodium chloride). The injection will be provided by the same maxillofacial surgeon. The participants are asked to clench their teeth to determine the site of the most intense muscle activity in the masseter and temporal muscles with palpation. Intramuscular BTX-A injections are administered on both sides at the location of the most intense muscle activity of the masseter (80 units) and temporalis (20 units). This technique is similar to other studies using BTX-A for the masseter and temporal muscles (Von Lindern et al., 2003; Guarda-Nardini et al., 2012; De la Torre Canales et al., 2021)

Description of measuring instruments and questionnaires Visual Analogue Scale (VAS) The VAS will be used to measure pain intensity. The VAS consists of a 100 mm line, with two set points, 0 (indicating no pain) and 10 (indicating worst imaginable pain). The participants rate their current pain by placing a mark on the line. Data are classified as metric. The test-retest reliability is good to excellent, with intraclass correlation coefficients (ICC's) ranging from 0.71 to 0.99 (Kahl & Cleland, 2005). In comparison with the numeric pain rating scale the VAS has up to 0.95 convergent validity (Kahl & Cleland, 2005). A study by Emshoff et al. (2010) showed an estimated minimal clinical difference of 19,5 mm in chronic TMD-related pain.

Oral health-related quality of life evaluation (OHIP-14) The OHIP-14 questionnaire is used to assess oral health-related quality of life on seven subscales. Every subscale includes two items. The subscales are: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and social handicap. The answer options are on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score ranges from 0 to 56 (metric), with a higher score indicating a more negative outcome. The test-retest reliability is moderate to high, with ICC's ranging from 0.78 to 0.90 (Van der Meulen et al., 2008). The smallest detectable difference (SDD) in dental disorders is measured at 5 points (Locker et al., 2004).

Mandibular Function Impairment Questionnaire (MFIQ) Mandibular function is assessed by the sum score of 17- item Dutch translation of the MFIQ (Kropmans et al., 1999). Each item is scored on a 5-point Likert scale with 0 indicating no difficulty and 4 being extremely difficult to perform a mandibular task, resulting in a total score ranging from 0 to 68 (metric). A higher score indicates higher levels of functional impairment. The test-retest reliability is moderate to high, with ICC's ranging from 0.69 to 0.96. The SDD is 10 points (Kropmans et al., 1999).

Maximal mouth opening Maximal mouth opening is measured at the distance between the incisal edges of the central incisors in millimeters. The measurement will be conducted with a metal ruler unassisted for the active mouth opening (AMO) as well as assisted for the passive mouth opening (PMO) according to the Dutch translation of the DC/TMD (Schiffman et al., 2014). Intra-rater reliability varied from 0.70 to 0.99. Interrater reliability varied from 0.90 to 1.00 (Walker et al., 2000). The mean of three measurements was used. The SDD in patients with painful restriction of the TMJ is 3 mm (Kropmans et al., 1999).

All outcome measures are assessed prior to the BTX injection (T0) and re-assessed at one (T1), three months (T2) and six months (T3) post-treatment by the same researcher. The researcher was external from the department of OMS and was not involved in any treatment session or treatment contact. All measurements are conducted without the presence of the healthcare practitioner providing the injections to avoid observer bias due to the patient-doctor relation. At all post treatment measurements, participants are asked if they had other treatments for their TMD-related myalgia and the exclusion criteria were reevaluated.

ELIGIBILITY:
Inclusion Criteria:

* TMD-related myalgia in accordance with the DC/TMD;
* Accepted BTX-A injections as treatment;
* Age ≥ 18 years;
* Understanding of the Dutch language to fill in the questionnaires.

Exclusion Criteria:

* Systemic inflammatory and connective tissue diseases (e.g., rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis);
* Surgery in the TMJ area < 12 months ago;
* Pain of dental origin;
* Limited cognitive functioning (not allowed to make medical decisions);
* Use of muscle relaxants, or aminoglycoside antibiotics;
* A history of allergic reactions to BTX;
* Pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study were adults with TMD-related myalgia according to the DC/TMD treated with a BTX-A injection. All participants were recruited at the department of Oral and Maxillofacial Surgery (OMS) of the Diakonessenhuis, Utrecht, The Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean pain rated with the VAS at 1, 3 and 6 months | Baseline, 1, 3 and 6 months
  The VAS will be used to measure pain intensity. The VAS consists of a 100 mm line, with two set points, 0 (indicating no pain) and 10 (indicating worst imaginable pain).

SECONDARY OUTCOMES:
Change from baseline in the mean oral health related quality of life rated with the OHIP-14 at 1, 3 and 6 months | Baseline, 1, 3 and 6 months
  The OHIP-14 questionnaire will be used to assess oral health-related quality of life on seven subscales. Every subscale includes two items. The subscales are: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and social handicap. The answer options are on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score ranges from 0 to 56 (metric), with a higher score indicating a more negative outcome.
Change from baseline in mean mandibular function rated by the MFIQ at 1, 3, and 6 months | Baseline, 1, 3 and 6 months
  Mandibular function will be assessed using the sum score of 17- item Dutch translation of the MFIQ (Kropmans et al., 1999). Each item is scored on a 5-point Likert scale with 0 indicating no difficulty and 4 being extremely difficult to perform a mandibular task, resulting in a total score ranging from 0 to 68 (metric). A higher score indicates higher levels of functional impairment.
Change from baseline in the mean maximal active and passive mouth opening at 1, 3 and 6 months | Baseline, 1, 3 and 6 months
  Maximal mouth opening will be measured at the distance between the incisal edges of the central incisors in millimeters. The measurements are conducted with a metal ruler unassisted for the active mouth opening (AMO) as well as assisted for the passive mouth opening (PMO) according to the Dutch translation of the DC/TMD .

CONTACTS AND LOCATIONS:
Overall Officials: Maurits HT de Ruiter, Dr., Study Director — Diakonessenhuis, Utrecht
Locations (1):
- Diakonessenhuis Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patel J, Cardoso JA, Mehta S. A systematic review of botulinum toxin in the management of patients with temporomandibular disorders and bruxism. Br Dent J. 2019 May;226(9):667-672. doi: 10.1038/s41415-019-0257-z. PMID 31076698
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Gil-Martinez A, Paris-Alemany A, Lopez-de-Uralde-Villanueva I, La Touche R. Management of pain in patients with temporomandibular disorder (TMD): challenges and solutions. J Pain Res. 2018 Mar 16;11:571-587. doi: 10.2147/JPR.S127950. eCollection 2018. PMID 29588615
- [Background] De la Torre Canales G, Poluha RL, Lora VM, Araujo Oliveira Ferreira DM, Stuginski-Barbosa J, Bonjardim LR, Cury AADB, Conti PCR. Botulinum toxin type A applications for masticatory myofascial pain and trigeminal neuralgia: what is the evidence regarding adverse effects? Clin Oral Investig. 2019 Sep;23(9):3411-3421. doi: 10.1007/s00784-019-03026-4. Epub 2019 Jul 24. PMID 31342244
- [Background] Chisnoiu AM, Picos AM, Popa S, Chisnoiu PD, Lascu L, Picos A, Chisnoiu R. Factors involved in the etiology of temporomandibular disorders - a literature review. Clujul Med. 2015;88(4):473-8. doi: 10.15386/cjmed-485. Epub 2015 Nov 15. PMID 26732121
- [Background] Sipahi Calis A, Colakoglu Z, Gunbay S. The use of botulinum toxin-a in the treatment of muscular temporomandibular joint disorders. J Stomatol Oral Maxillofac Surg. 2019 Sep;120(4):322-325. doi: 10.1016/j.jormas.2019.02.015. Epub 2019 Feb 23. PMID 30807862